CLINICAL TRIAL: NCT00589628
Title: Multi Center Prospective Registry of Infliximab Use for Childhood Uveitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Egla C. Rabinovich (Other)
Collaborators: Childhood Arthritis and Rheumatology Research Alliance (Other)
Responsible Party: Sponsor-Investigator, Egla C. Rabinovich, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000057
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Uveitis
Keywords: Childhood; Uveitis
MeSH Terms: conditions — Uveitis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 5mg/kg/dose of infliximab IV every 4 weeks for 9 doses
  Interventions: Drug: infliximab
- 2 (Active Comparator): 10mg/kg/dose of infliximab IV every 4 weeks for 9 doses.
  Interventions: Drug: infliximab

INTERVENTIONS:
Drug: infliximab — 5mg/kg/dose IV at 4 week intervals
  Other Names: Remicade
  Arms: 1
Drug: infliximab — 10mg/kg/dose IV at 4 week intervals
  Other Names: Remicade
  Arms: 2

SUMMARY:
The primary objective of this study is to examine the efficacy of infliximab for the treatment of persistent uveitis in children. Participants (4-18 years of age) will be randomly assigned to either 5mg/kg or 10mg/kg dose of infliximab to be administered by intravenous infusion at four week intervals. Participant responses will be measured at at four to eight week intervals for up to ten months.

DETAILED DESCRIPTION:
Pediatric rheumatologists often use infliximab in the treatment of childhood uveitis, at this time there are no prospective studies for this use. Participants will be randomized to initial suggested dose of infliximab (5 mg/kg/dose vs 10 mg/kg/dose) and data will be collected prospectively with regard to ophthalmologic outcomes. Study participants will be followed for up to 10 months to determine efficacy and side effects, and an additional 30 days for safety reports. Descriptive statistics will be gathered on participant demographics, uveitis characteristics, change in immunosuppressive medications, number of responders, ophthalmologic measures and change in corticosteroid dose during the study period. Initial to final dose will be examined by paired t-test. The proportion of responders in the 5 mg/kg initial dose group will be compared to the 10 mg/kg/dose by a Chi-square or Fisher's exact test, depending on numbers available. Predictors of response will be examined by logistic regression.

ELIGIBILITY:
Inclusion Criteria:.

1. Ages 4 to 18 years old,
2. Non-infectious uveitis
3. Persistent uveitis uncontrolled by topical medications, or unacceptable side effects of topical medications.
4. Failure of at least six weeks of treatment with a non-biological disease modifying agent such as methotrexate, cyclosporine, mycophenolate mofetil, or azathioprine.
5. Ability to provide informed consent (subject or parent/guardian)
6. Onset of uveitis < 16 years of age.
7. Topical ophthalmologic treatments allowed.
8. Systemic corticosteroid use at entry may be allowed.
9. Willingness to use acceptable contraception if sexually active for the duration of the study and for 6 months after receiving the last infliximab infusion.
10. Concomitant methotrexate must be taken at time of initiation of infliximab
11. Participant must be able to cooperate for a non-sedated slit lamp exam and visual acuity examination.
12. Negative Purified Protein Derivative (PPD) placed and read within 1 month of initiation of infliximab
13. The screening laboratory test results must meet the following criteria:

    * WBC (white blood cell count): within normal range for institution
    * ANC (absolute neutrophil count): within normal range for institution
    * Hemoglobin: greater than 10 grams/deciliter
    * Platelets: within normal range for institution
    * Serum Creatinine: within normal range for age
    * AST - aspartate aminotransferase - within normal range for institution
    * ALT - alanine aminotransferase- within normal range for institution

Exclusion Criteria:

1. Previous use of biologic medications for uveitis.
2. Intraocular steroid injection or ophthalmologic surgery within the preceding 3 months.
3. Uveitis due to trauma or intraocular surgery
4. Females who are pregnant, nursing, or planning pregnancy within 6 months after the last infliximab infusion.
5. Males who plan on fathering a child within 6 months after their last infliximab infusion.
6. A history of a known allergy to murine products.
7. Documentation of seropositivity for human immunodeficiency virus (HIV).
8. Documentation of a positive test for hepatitis B surface antigen or hepatitis C
9. A known history of a serious infection (e.g., hepatitis, pneumonia, or pyelonephritis) in the previous 3 months.
10. An opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening.
11. A concomitant diagnosis or history of congestive heart failure.
12. A history of lymphoproliferative disease.
13. Any known malignancy or a history of malignancy.
14. Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
15. Use of any investigational drug within 30 days prior to screening or within five half-lives of the first dose of the investigational agent, whichever is longer.
16. Presence of a transplanted solid organ.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Egla Rabinovich, MD. MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Heiligenhaus A, Foeldvari I, Edelsten C, Smith JR, Saurenmann RK, Bodaghi B, de Boer J, Graham E, Anton J, Kotaniemi K, Mackensen F, Minden K, Nielsen S, Rabinovich EC, Ramanan AV, Strand V; Multinational Interdisciplinary Working Group for Uveitis in Childhood. Proposed outcome measures for prospective clinical trials in juvenile idiopathic arthritis-associated uveitis: a consensus effort from the multinational interdisciplinary working group for uveitis in childhood. Arthritis Care Res (Hoboken). 2012 Sep;64(9):1365-72. doi: 10.1002/acr.21674. PMID 22438273
- [Background] Ardoin SP, Kredich D, Rabinovich E, Schanberg LE, Jaffe GJ. Infliximab to treat chronic noninfectious uveitis in children: retrospective case series with long-term follow-up. Am J Ophthalmol. 2007 Dec;144(6):844-849. doi: 10.1016/j.ajo.2007.08.018. Epub 2007 Oct 22. PMID 17953940
- [Result] Saurenmann RK, Levin AV, Rose JB, Parker S, Rabinovitch T, Tyrrell PN, Feldman BM, Laxer RM, Schneider R, Silverman ED. Tumour necrosis factor alpha inhibitors in the treatment of childhood uveitis. Rheumatology (Oxford). 2006 Aug;45(8):982-9. doi: 10.1093/rheumatology/kel030. Epub 2006 Feb 3. PMID 16461435
- [Result] Kahn P, Weiss M, Imundo LF, Levy DM. Favorable response to high-dose infliximab for refractory childhood uveitis. Ophthalmology. 2006 May;113(5):860-4.e2. doi: 10.1016/j.ophtha.2006.01.005. Epub 2006 Mar 20. PMID 16545455
- [Result] Rajaraman RT, Kimura Y, Li S, Haines K, Chu DS. Retrospective case review of pediatric patients with uveitis treated with infliximab. Ophthalmology. 2006 Feb;113(2):308-14. doi: 10.1016/j.ophtha.2005.09.037. Epub 2006 Jan 10. PMID 16406545
- See also: Research Information. Click on current studies — http://carragroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab 5 mg/kg: 5mg/kg/does of infliximab IV at 4 week intervals
- Infliximab 10 mg/kg: 10mg/kg/dose of infliximab Iv at 4 week intervals
Period: Overall Study
Arm/Group | Infliximab 5 mg/kg | Infliximab 10 mg/kg
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 5 mg/kg of Infliximab: 5mg/kg/does of infliximab IV at 4 week intervals
- 10 mg/kg of Infliximab: 10mg/kg/dose of infliximab Iv at 4 week intervals
- Total: Total of all reporting groups
Arm/Group | 5 mg/kg of Infliximab | 10 mg/kg of Infliximab | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 13
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Effects of Infliximab on Uveitis Disease Activity.
Description: Number of subjects with improvement in uveitis, defined as a two step decrease in level of inflammation (as defined by SUN criteria, AC cells, vitreous haze) or decrease to grade 0. A grading scheme of 0 indicating (<1 cell/ocular field) low levels of inflammation to 4+ indicating (>50 cells/ocular field) indicating high levels of inflammation.
Time Frame: 9 months
Population: 1 subject lost to follow up
Measure: Number; unit: participants
Groups:
- Infliximab 5mg/kg: 5mg/kg/does of infliximab IV at 4 week intervals
- Infliximab 10mg/kg: 10mg/kg/dose of infliximab Iv at 4 week intervals
Arm/Group | Infliximab 5mg/kg | Infliximab 10mg/kg
Number analyzed (Participants) | 7 | 6
participants | 3 [0 to 4] | 6 [0 to 4]

ADVERSE EVENTS:
Arm/Group | 5 mg/kg of Infliximab | 10 mg/kg of Infliximab
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/6
Other Adverse Events (participants affected / at risk) | 2/7 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg/kg of Infliximab (N=7) | 10 mg/kg of Infliximab (N=6)
Fever (Infections and infestations) | 0 (0) | 1 (1) — Hospitalization for a positive blood culture, but repeat negative and felt to be consistent with a contaminated culture. Subject also had myalgias and ear cellulitis. Refused further follow up
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg/kg of Infliximab (N=7) | 10 mg/kg of Infliximab (N=6)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fever blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study recruitment was difficult and slow. Optimal number not achieved in this descriptive study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No